CLINICAL TRIAL: NCT03869476
Title: Pilot Study for the Development of a Non-invasive Diagnostic Score to Differentiate Between Essential Thrombocythemia, Premyelofibrosis and Myelofibrosis
Brief Title: Pilot Study for the Development of a Diagnostic Score to Differentiate Myeloproliferative Neoplasms.
Acronym: BioScoreSMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 49RC18_0153_1
Record Dates: First submitted 2019-03-06; First posted 2019-03-11 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Myeloproliferative Disorder; Essential Thrombocythemia; Primary Myelofibrosis, Prefibrotic Stage; Primary Myelofibrosis, Fibrotic Stage
MeSH Terms: conditions — Myeloproliferative Disorders; Thrombocythemia, Essential; Primary Myelofibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BioscoreSMP cohort (Experimental)
  Interventions: Diagnostic Test: Non-invasive diagnosis score

INTERVENTIONS:
Diagnostic Test: Non-invasive diagnosis score — * spleen fibrosis by elastography
  * plasma cytokines levels
  * mutationnal landscape by NGS
  * CD34 circulating cells

SUMMARY:
Prospective study for the development of a non-invasive score for differentiating prefibrotic myelofibrosis from essential thrombocytosis and overt myelofibrosis.

DETAILED DESCRIPTION:
The diagnostic criteria for myeloproliferative neoplasia have recently been revised in the WHO 2016 classification, which now recognizes a new entity between essential thrombocythemia (TE) and overt myelofibrosis (or primary myelofibrosis): prefibrotic myelofibrosis. Prefibrotic myelofibrosis patients seem to have a poorer prognosis compared to essential thrombocythemia in term of overall survival and myelofibrotic evolution. The dichotomy between these diseases is based on the bone marrow biopsy evaluation and is challenging with a lack of reproducibility showed in the literature.

This study aims to develop a diagnostic non-invasive score for differentiating prefibrotic myelofibrosis from essential thrombocytosis and overt myelofibrosis.

The parameters studied are :

* spleen fibrosis by elastography
* plasma cytokines levels
* mutationnal landscape by NGS
* CD34 circulating cells

Bone marrow biopsy were reviewed by 2 anatomopathologists. Number of patients to be enrolled : 130

ELIGIBILITY:
Inclusion Criteria:

* Adult (18 years of age or older) with the diagnosis of essential thrombocytosis, prefibrotic myelofibrosis or overt myelofibrosis according to WHO 2016 criteria;
* Patient who has not received specific treatment for neoplasms;
* Patient who has signed the consent to participate in the study;
* Patient who has consented to be included in the "Malignant Haemopathies" collection at the University Hospital of Angers or Brest and for whom the samples necessary for the study are available in the biocollection.

Exclusion Criteria:

* Patient with another hematologic neoplasm or progressive cancer at the time of diagnosis;
* Patient with a diagnosis of secondary myelofibrosis;
* Pregnant or breastfeeding woman;
* Person prived of liberty by judicial or administrative decision;
* Person subject to a legal protection measure;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2019-07-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
WHO 2016 criteria for prefibrotic myelofibrosis, essential thrombocytosis and overt myelofibrosis diagnosis | At the time of diagnosis : disease classification
  Assessment of the non-invasive diagnostic score against the WHO diagnosis

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Chu Angers, Angers
  - CHRU de Brest - Hôpital Morvan, Brest

IPD SHARING:
Plan to Share IPD: Yes
Data of study protocol, Statiscal analysis plan and the infromed consent form will be made available after the study completion
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available within 1 year of study completion
Access Criteria: Data access requests will be reviewed and requestors will be required to sign a data acess agreement